CLINICAL TRIAL: NCT00854269
Title: Screening and Identification of Novel Diagnostic and Prognosis Biomarkers on Cervical Cancers
Brief Title: Screening and Identification of Biomarkers on Cervical Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chi-An Chen/Professor, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200705075R
Record Dates: First submitted 2008-04-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: surgery — cervical biopsy or specimen of hysterectomy

SUMMARY:
Cervical cancer the most frequent neoplasm and the fifth mortality rate of malignancies of the women in the world. It results in about 1,000 women in Taiwan and about 200,000 women worldwide dying of cervical cancer each year. Human papilloma viruses (HPV) have been consistently implicated in causing cervical cancer especially those high-risk types (HPV 16,18,31,45) have been strongly associated with cervical cancer. Around 50-80 % of women are infected by HPV within their whole lives. However, only 1% of HPV-infected women have cervical cancer eventually. Seventy and 91% of HPV infection could be cleaned up by host immune responses within 1 and 2 years later. It shows that host immunity plays an important role in the progression, persistence, or regression of HPV infection.

There are two main defense lines in the host immunity including innate immunity and adoptive immunity. Adoptive immunity plays more important roles in the defense of HPV infections than innate immunity. The adoptive immunity could be further divided into humoral immunity and cell-mediated immunity. Humoral immunity regulated by Th2 helper T lymphocytes to generate memory B cells to produce antibody which provide the protective function to HPV infection. Cell-mediated immunity regulated by Th1 helper T lymphocytes to induce antigen-specific cytotoxic T cells which could kill the HPV-infected cells. Although there are many researches focused on the immunity to HPV infection, there is no conclusion about the relationship between humoral and cell-mediated immunities on HPV infection and roles of humoral and cell-mediated immunities in the prognosis of HPV-infected population and cervical cancer patients.

Our research team has focused on the establishment of platforms on cell-mediated immunity to HPV infection and on the correlation of cell-mediated immunity and prognosis of HPV-infected population and cervical cancer patients for years. In order to survey the host immunity to HPV infection more comprehensively, we propose this 3-year proposal. First, we would like to set up the platforms to survey the humoral immunity to HPV infection in normal population and patients with CIN lesion or cervical cancer. Second, we would to elucidate the correlation between humoral immunity and status and clinico-pathologic items of HPV-infected populations. Third, we would like to survey if the humoral immunity correlate with the prognosis of patients with cervical lesions. Fourth, we would like to elucidate the correlation betweenHLA haplotype and humoral immunity in HPV-infected populations. Our research results will have a more comprehensive overview in the host immunity to HPV infection and its related diseases. It could provide more information in the prevention and treatment of HPV infection in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* People infected with HPV type 16 but without CIN lesions
* Patients with CIN lesions
* Patients with cervical cancer from National Taiwan University Hospital
* Informed consent is obtained, and the protocols are reviewed and approved by the appropriate Investigative Review Boards.

Exclusion Criteria:

* None

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-05 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | from disease diagnosis to death

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan